CLINICAL TRIAL: NCT02090257
Title: Pediatric Heart Transplantation: Transitioning to Adult Care
Acronym: TRANSIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Elfriede Pahl, MD, Attending Physician, Division of Cardiology, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1R34HL111492 (NIH)
Record Dates: First submitted 2014-03-05; First posted 2014-03-18 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Heart Transplantation
Keywords: Heart transplant recipients who are entering into adult care.

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TRANSIT, behavioral (Experimental): The intervention group will receive more guidance during their transition from a pediatric center to the adult center
  Interventions: Behavioral: TRANSIT
- Usual Care Group (No Intervention): The usual care group will receive a standard transfer of care from a pediatric center to an adult center.

INTERVENTIONS:
Behavioral: TRANSIT — Educational Modules, staff follow up.
  Arms: TRANSIT, behavioral

SUMMARY:
The purpose of this pilot trial, Transitioning to Adult Care (TRANSIT), is to develop and test an intervention (i.e., a standardized, tailored transition program focused on enhancing adherence) to improve outcomes for emerging adults who underwent heart transplantation as children and transfer to adult care.

ELIGIBILITY:
Inclusion Criteria:

* Have received a heart transplant at a children's hospital and are ready to transition, as determined by the pediatric heart transplant cardiologist, to the adult heart transplant center with whom a collaborative relationship has been established;
* 18 years or older;
* Able to speak, read at a fifth grade level or above, and write English;
* Physically able to participate.

Exclusion Criteria:

* History of psychiatric hospitalization within the last 3 months, assessed on a case-by-case basis with exclusion only if patients could not potentially benefit from the intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
To assess the feasibility of TRANSIT by measuring the transition program adherence for those randomized to the intervention and survey completion for all participants. | 6 months
  Investigators hypothesize that by the end of the 3 month transition program and 6 months of follow-up, 84% of patients will be retained; 80% will participate in the program (module completion, discussion, and follow-up); and 100% will complete at least 80% of the survey instruments at each data collection point.

SECONDARY OUTCOMES:
To determine the efficacy of TRANSIT on patient-level outcomes . | 6 months
  The following patient level outcomes will be measured:
  1. At 3 months post intervention and 6 months follow-up, emerging adult heart transplant recipients who participate in TRANSIT will have lower CNI SD (i.e., SD <2.5 for tacrolimus and cyclosporine), than patients who receive usual care.
  2. At 3 months post intervention and 6 months follow-up, emerging adult heart transplant recipients who participate in TRANSIT will have a higher percentage of CNI levels within the target range (i.e., < 50% of CNI blood levels out of target range for individual patients as reported by their transplant center), better self-reported adherence to the medical regimen, and fewer episodes of treated acute rejection, than patients who receive usual care.
  3. At 3 months post intervention and 6 months follow-up, emerging adult heart transplant recipients who participate in TRANSIT then patients who receive usual care.
To determine the efficacy of TRANSIT on meso-level outcomes. | 6 Months
  These will be measured based on the use of health care resources: rates of appointments for clinic and CNI blood draws and number of all-cause days re-hospitalized

CONTACTS AND LOCATIONS:
Overall Officials: Elfriede Pahl, MD, Principal Investigator — Ann and Robert Lurie Children's Hospital; Kathleen Grady, PhD, Principal Investigator — Northwestern University
Locations (6):
- United States (6):
  - Loma Linda University, Loma Linda, California
  - Universtiy of Colorado Denver/Children Colorado, Aurora, Colorado
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Columbia University, New York, New York
  - Children's Hospital of Philadelphia/University of Pennsylvania, Philadelphia, Pennsylvania